CLINICAL TRIAL: NCT02609217
Title: Parents' Expectations and Experiences Around Cesarean Section in Belgium
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Tim Van Mieghem, Assistant professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: 58593
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cesarean Section
Keywords: elective; cesarean
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiparous: 12 multiparous women and their partners, planned to undergo elective term cesarean section.
  Interventions: Other: Questionnaires and interviews
- Nulliparous: 12 nulliparous women and their partners, planned to undergo elective term cesarean section.
  Interventions: Other: Questionnaires and interviews

INTERVENTIONS:
Other: Questionnaires and interviews

SUMMARY:
The aim of this study is to gain insight in the experiences and expectations of Belgian parents concerning primary cesarean section. This will be achieved by structured patient interviews and questionnaires in 24 women undergoing the procedure and their partners. This group will be divided into two subgroups of 12 multiparous and 12 nulliparous women and their partners.

DETAILED DESCRIPTION:
The subjects in both groups will be interviewed twice and will receive three questionnaires. One to two weeks prior to the scheduled cesarean section and during a scheduled obstetric outpatient visit, the first interview and questionnaire will be administered to the couple. A second questionnaire will be provided while still hospitalized (5 days post partum), to both mother and partner. Six weeks post partum, during a scheduled obstetric outpatient visit, the couple will be interviewed for the last time and will be asked to complete the third and last questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Partner available
* 18-50 years of age
* Singleton pregnancy
* Booked for planned cesarean section ≥37 weeks of gestation
* Dutch-speaking
* Informed consent given

Exclusion Criteria:

* Emergency cesarean section
* <18 years of age or >50 years of age
* Multiple pregnancy
* Inability to provide consent (language, etc.)
* Partner not consenting
* BMI >35 kg/m2
* Maternal or fetal pathologies expected to affect pre and postnatal maternal/neonatal management

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women planned to undergo term elective cesarean section selected from antenatal low-risk clinic.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Information on parents' fears and expectations around cesarean section | 6 weeks post partum
  Information on parents' fears and expectations around cesarean section will be obtained using structured patient interviews and questionnaires.

SECONDARY OUTCOMES:
Quantitative data on postoperative pain after cesarean section | 6 weeks post partum
  Quantitative data on postoperative pain after cesarean section will be obtained using VAS (Visual Analogue Scale) pain scores.
Data on the experience of postoperative pain after cesarean section | 6 weeks postpartum
  Data on the experience of postoperative pain after cesarean section will be obtained by content analysis of structured interviews.
Data on frequency of breastfeeding after cesarean section | 6 weeks postpartum
  Frequency of breastfeeding after cesarean section will be described by number of breastfeeds per 24h.
Qualitative data of breastfeeding after cesarean section | 6 weeks postpartum
  Data on quality of breastfeeding after cesarean section will be obtained using LATCH breastfeeding scores.
Data on the experience of breastfeeding after cesarean section | 6 weeks postpartum
  Data on the experience of breastfeeding after cesarean section will be obtained by content analysis of structured interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium